CLINICAL TRIAL: NCT06081088
Title: The Effectiveness of Graded Motor Imagery Training in Patients With Shoulder Impingement Syndrome
Brief Title: Graded Motor Imagery Training in Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Marmara Uni.
Record Dates: First submitted 2023-10-02; First posted 2023-10-12 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Impingement Syndrome; Pain
Keywords: Shoulder Impingement Syndrome; Mirror Neurons; Pain; Functional Status; Rehabilitation
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Study group: "Graded Motor Imagery Training + Conventional Physiotherapy"
  In this group, each participant will be received a treatment protocol consisting of Graded Motor Imagery training, conventional physiotherapy, and home exercises.
  * Graded Motor Imagery (GMI)
  * Conventional Physiotherapy Program
  * Home Exercise Program
  Interventions: Other: Graded Motor Imagery (GMI) training; Other: Conventional Physiotherapy; Other: Home Exercise Program
- Group 2 (Active Comparator): Control group: "Conventional Physiotherapy"
  In this group, each participant will be received a treatment protocol consisting of conventional physiotherapy, and home exercises.
  * Conventional Physiotherapy Program
  * Home Exercise Program
  Interventions: Other: Conventional Physiotherapy; Other: Home Exercise Program

INTERVENTIONS:
Other: Graded Motor Imagery (GMI) training — GMI consists of three basic components:
  1. Left / Right Discrimination training (Lateralization training): For lateralization training, patients will be trained by asking them to distinguish between right and left with images taken at various angles and positions in the RecogniseTM (NOI-Australia) applications (shoulder and hand sections) (In weeks 1 and 2).
  2. Motor Imagery (Explicit Motor Imagery): At this stage, the participant will be asked to imagine doing various functional activities (brushing teeth, combing hair, etc.) in the position they feel most comfortable in and in a quiet environment (In weeks 2 and 3).
  3. Mirror Therapy (providing visual feedback through a mirror): In this phase, active ROM exercises and progressive resistance exercises with simultaneous movement of the affected and unaffected extremities will be applied using a standard size posture mirror (In weeks 3-6).
  This program will be applied for 6 weeks (3 sessions per week).
  Arms: Group 1
Other: Conventional Physiotherapy — Conventional physiotherapy program includes passive, active-assistive (wand exercises) and active ROM exercises for shoulder joint, passive / active posterior and anterior capsule stretching exercises, superior-inferior, mediolateral and distraction techniques for scapular mobilization exercises, shoulder flexion, abduction, internal and external rotation muscles strengthening exercises, static and dynamic stabilization exercises for proprioception exercises. To reduce the pain that may occur after exercises, cold application and Transcutaneous Electrical Nerve Stimulation (TENS) will be applied to benefit from their analgesic effects. Cold application will be applied around the shoulder using a coldpack (gel pack) cold therapy for 15 minutes. Conventional TENS application around shoulder will be performed using a TENS device and four separate 2 × 2 inch self-adhesive electrodes for 15 minutes.This program will be applied for 6 weeks (3 sessions per week).
Other: Home Exercise Program — The home exercises program includes shoulder jonit active ROM exercises, active posterior and anterior shoulder capsule stretching exercises, shoulder flexion, abduction, internal and external rotation muscles strengthening exercises, shoulder proprioception exercises, and cold therapy. This program will be applied for 6 weeks (3 sessions per week).

SUMMARY:
The aim of this study is to investigate the effects of Graded Motor Imagery (GMI) training on pain, functionality, disability and daily living activities in patients diagnosed with Shoulder Impingement Syndrome.

DETAILED DESCRIPTION:
In this study 42 voluntary patients with Shoulder Impingement Syndrome, aged between 25-65 years will be randomly divided into two groups; group1: "GMI + Conventional Physiotherapy", group 2: "Conventional Physiotherapy".

All participants will receive treatment with a physiotherapist three times a week for six-weeks (18 sessions). At the end of the 6th week, it will be followed regularly with a six-week home exercise program. It will be evaluated by a physiotherapist three times in total (before treatment, at the end of six-weeks of treatment and after six-weeks of follow-up). In addition, all patients will undergo an interim evaluation in terms of primary outcome measures (VAS and DASH score) at week three. The shoulder pain on activity, at rest and at night will be assessed with Visual Analog Scale (VAS), Joint Range of Motion (ROM) will be measured with digital goniometer, strength of shoulder flexor, abductor, external and internal rotator muscles will be assessed with digital dynamometer, functional status will be evaluated with Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, functional status of the hand will be evaluated with Jebsen-Taylor Hand Function Test (JTHFT), lateralization evaluation will be assessed with the Recognise™ application (Shoulder and Hand), and motor imagery will be evaluated with the Kinesthetic and Visual Imagery Questionnair (KVIQ). Patient satisfaction will be evaluated by the Global Rating of Change scale.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 25-65 years old,
* Having been diagnosed with Shoulder Impingement Syndrome by physical examination and MRI as a result of shoulder pain lasting at least 3 months,
* Presence of a painful arc between 60° and 120° in shoulder flexion / abduction (elevation) movements,
* The Standardized Mini Mental Test result must be at least 24 points,
* Not having seen imagery practice before,

Exclusion Criteria:

* Having severe mental and communication problems,
* Having undergone surgical treatment on the same upper extremity,
* Presence of acute trauma, peripheral nervous system lesion, fracture or complete tendon rupture in the affected shoulder,
* Presence of other pathologies such as adhesive capsulitis of the shoulder joint complex and glenohumeral instability,
* Presence of radiotherapy history on the same side as the affected shoulder,
* Presence of congenital deformity,
* Symptomatic cervical spine pathology,
* Presence of other neurological or rheumatological disorders affecting upper motor function,
* Having any chronic disease that would prevent participation in the treatment program,
* Having attended a physiotherapy program within the last month.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline, Interim evaluation (At the end of the 3rd week), After the six-week intervention, After six-weeks of follow-up
  Pain intensity will be assessed with Visual Analog Scale (VAS). The VAS is usually a horizontal line, 10 cm in length, anchored by word descriptors at each end with "No Pain" (score of zero) on the left side up to "pain as bad as it could be" or the "worst imaginable pain" (Score of 100 [100-mm scale]) on the right side.The patient will be asked to mark the line point that represented his or her current pain.
Functional Status | Baseline, Interim evaluation (At the end of the 3rd week), After the six-week intervention, After six-weeks of follow-up
  The disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used in shoulder functional status evaluation. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. 21 of the questions of the survey question the ability to perform functional activities, 5 question the pain, and 4 question the psychosocial effects of the disease. Each question is scored using a 5-point Likert scale ranging from 1 to 5 (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not at all). Higher scores indicate better functional status.

SECONDARY OUTCOMES:
Active Range Of Motion (AROM) | Baseline, After the six-week intervention, After six-weeks of follow-up
  A digital goniometer will be used to measure shoulder active joint range of motion. While the patient is lying in the supine position, shoulder active flexion, active abduction, and then shoulder internal (internal) and external (external) rotation ROM measurements will be made with the shoulder in 90 degrees abduction and the elbow in 90 degrees flexion.
Isometric Muscle Strength | Baseline, After the six-week intervention, After six-weeks of follow-up
  Isometric muscle strength of shoulder flexor, abductor, external and internal rotator muscles will be evaluated with a hand-held dynamometer. During muscle strength evaluation, patients will be asked to perform maximal voluntary isometric contraction while in a sitting position. Measurements will be repeated 3 times (5 seconds of contraction followed by 30 seconds of rest) for the affected side and the average of the 3 measurements will be taken and the resulting value will be recorded in kilograms (kg).
Functional Status Of the Hand | Baseline, After the six-week intervention, After six-weeks of follow-up
  Jebsen-Taylor Hand Function Test (JTHFT) will be used to evaluate the functional status of the hand. JTHFT is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living. The JTHFT has seven subsets which are writing, simulated page-turning, lifting small objects, simulated feeding, stacking, and lifting large, lightweight, and heavy objects. Time will be recorded in this test. Except for writing, other tasks are done separately with both hands. The completion time of the tasks refers to the subtask scores and total score of JTHFT. The total score is obtained by adding up the completion time of the six tasks other than writing for the dominant and non-dominant hands.
Left/right discrimination (Lateralization) | Baseline, After the six-week intervention, After six-weeks of follow-up
  Right-Left Discrimination will be evaluated with Recognise™ applications (Shoulder and Hand) developed by the "Neuro Orthopedic Institute".
Kinesthetic and Visual Imagery Questionnaire (KVIQ) | Baseline, After the six-week intervention, After six-weeks of follow-up
  Motor imagery ability will be assessed with the Kinesthetic and Visual Imagery Questionnaire (KVIQ). The participant gives a score between 1 and 5 for the image he/she imagines: "1 point: no image, 5 points: as clear as the original." This process is repeated for each task and at the end of the survey, kinesthetic imagery score, visual imagery score and total score are calculated.
Global Rating of Change scale (Patient Satisfaction) | After the six-week intervention
  Patient satisfaction regarding improvement in shoulder function will be evulated by the Global Rating of Change scale. All participants will be asked to rate their condition after a six-week intervention period compared to baseline by indicating whether they have improved significantly, improved slightly, unchanged, deteriorated slightly, or deteriorated significantly in this study.

CONTACTS AND LOCATIONS:
Overall Officials: MASOUD AMIR RASHEDI BONAB, PhD, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Başıbüyük, Süreyyapaşa Başıbüyük Yolu Sk No:4/B, 34854 Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araya-Quintanilla F, Gutierrez-Espinoza H, Jesus Munoz-Yanez M, Rubio-Oyarzun D, Cavero-Redondo I, Martinez-Vizcaino V, Alvarez-Bueno C. The Short-term Effect of Graded Motor Imagery on the Affective Components of Pain in Subjects with Chronic Shoulder Pain Syndrome: Open-Label Single-Arm Prospective Study. Pain Med. 2020 Oct 1;21(10):2496-2501. doi: 10.1093/pm/pnz364. PMID 32003812
- [Background] Sawyer EE, McDevitt AW, Louw A, Puentedura EJ, Mintken PE. Use of Pain Neuroscience Education, Tactile Discrimination, and Graded Motor Imagery in an Individual With Frozen Shoulder. J Orthop Sports Phys Ther. 2018 Mar;48(3):174-184. doi: 10.2519/jospt.2018.7716. Epub 2017 Dec 19. PMID 29257926
- [Background] Louw A, Puentedura EJ, Reese D, Parker P, Miller T, Mintken PE. Immediate Effects of Mirror Therapy in Patients With Shoulder Pain and Decreased Range of Motion. Arch Phys Med Rehabil. 2017 Oct;98(10):1941-1947. doi: 10.1016/j.apmr.2017.03.031. Epub 2017 May 5. PMID 28483657
- [Background] Moseley GL. Graded motor imagery for pathologic pain: a randomized controlled trial. Neurology. 2006 Dec 26;67(12):2129-34. doi: 10.1212/01.wnl.0000249112.56935.32. Epub 2006 Nov 2. PMID 17082465